CLINICAL TRIAL: NCT06052215
Title: Effect of Online Information Cards Education on Women's Perception of Family Planning Disability, Attitudes and Behaviors in the Postpartum Period
Brief Title: Effect of Online Information Cards Education on Women's Perception of Family Planning Behaviors in the Postpartum Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, Ayse Cal, Assoc. Prof., Ankara Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: E-81477236-604.01.01-1927
Record Dates: First submitted 2023-09-07; First posted 2023-09-25 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Obstetric Care of the Giving Birth
Keywords: Family Planning; Health Education; Postpartum Period; Women; Nursing
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Solomon-1 (Experimental)
  Interventions: Behavioral: Online Information Cards Education
- Solomon-2 (Experimental): No pretest measurement
  Interventions: Behavioral: Online Information Cards Education
- Solomon-3 (No Intervention)
- Solomon-4 (No Intervention): No pretest measurement

INTERVENTIONS:
Behavioral: Online Information Cards Education — Providing family planning education to women through online information cards
  Arms: Solomon-1; Solomon-2

SUMMARY:
It is emphasized that the contraception knowledge of women in Turkey is insufficient and the rate of use of modern family planning methods should be increased. In this study, it is aimed to evaluate the effect of family planning education given via online information canrds on women's perception of disability, attitudes and behaviors in the postpartum period. The study is planned to be conducted in a randomized controlled experimental type using the Solomon four-group design. In the study, it is planned to make up a total of 150 women determined by using the G*Power program. The research will be carried out online with the women followed in Ankara Etlik City Hospital-Gynecology Hospital Obstetrics Clinics.

The data of the research will be collected with Introductory Information Form, Family Planning Method Usage History Form, Perception of Obstacles in Using Contraceptive Methods Scale and Family Planning Attitude Scale. The data will be analyzed using the SPSS 25.0 program. In the evaluation of the data; descriptive statistics, independent sample t-test, paired samples t-test, anova will be used.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization in Turkey Ankara Etlik City Hospital-Gynecology Hospital Obstetrics Clinics on the dates of the research
* Having had a cesarean or normal birth
* Being sexually active
* Being a woman aged 18 or over who has given birth
* Volunteering to participate in research
* Having the ability to read and understand Turkish
* Having a smart phone and internet access to access online information cards

Exclusion Criteria:

* Women with tubal ligation after cesarean section
* Women whose partner has had a vasectomy
* Women who received an Intrauterine Device at the time of delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2023-07-26 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Perception Scale of Barriers to Contraceptive Use | 1-3 mounth
  The lowest score that can be obtained from the scale is 31 and the highest score is 155. A high score from the scale indicates that the perceived barriers to the use of contraceptive methods are high.
Family Planning Attitude Scale | 1-3 mounth
  This scale, consisting of 34 items, is a five-point Likert type. The total score is obtained by adding the items in the scale, and a minimum of 34 and a maximum of 170 points can be obtained. An increase in the scale score indicates that family planning attitudes have changed positively.
The rate of use of family planning methods by women | 3. mounth
  Have you started using family planning methods? The question will be asked and the answer will be Yes or No.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Medipol University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No